CLINICAL TRIAL: NCT05513339
Title: Effect of Sleep Deprivation on Cognitive Function Among Cardiology Fellows
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Alexander Hajduczok, Principal Investigator, Thomas Jefferson University
Other Study IDs: 22D.689
Record Dates: First submitted 2022-08-18; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Wellness; Burnout; Sleep Deprivation; Executive Function
Keywords: WHOOP strap 4.0; Remote Monitoring
MeSH Terms: conditions — Burnout, Psychological; Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiology Fellows: Cardiology fellows at Thomas Jefferson University Hospital (PGY4-PGY6)
  Interventions: Device: WHOOP strap 4.0

INTERVENTIONS:
Device: WHOOP strap 4.0 — Subjects will wear the WHOOP strap 4.0 for continuous physiologic monitoring.

SUMMARY:
A reliable method for monitoring sleep, stress, and burnout among cardiology fellows is critically needed. To address this gap, our team aims to utilize the cost-effective WHOOP strap 4.0 wearable device to continuously capture stress-relevant physiologic data (i.e., sleep hours, heart rate variability, respiration rate, resting heart rate) among up to 21 Cardiology Fellows Thomas Jefferson University Hospital for 6 months.

DETAILED DESCRIPTION:
Conventional methods of qualifying personal wellbeing are limited by poor insight about the emotional and behavioral corollaries of stress and burnout (e.g., depersonalization, sleep alterations, heart rate variability). While self-care is often the preferred option for those coping with stress or burnout in challenging situations, it may be the only option in low-resource settings with limited access to professional management. Similarly, many healthcare workers and trainees acknowledge that self-care is a critical component to overall wellbeing, yet they also admit that multiple barriers interfere with the effectiveness of this practice. First, self-care interventions can only be effective if impacted persons recognize the need for interventions, act on that need, and learn which methods are effective on an individual basis. Furthermore, testing modalities (e.g., hormonal assays, polysomnography, electrophysiology) for stress and its downstream syndrome of burnout not only are prohibitively expensive, but they also require significant time and cannot be broadly disseminated within reasonable limits. As such, approaches for monitoring parameters of wellness are critically needed, and if successful, those data can allow for streamlined mental health interventions for those completing fellowship training before symptoms of burnout escalate further.

Aim 1: To determine whether physiologic metrics of sleep and heart rate variability correlate with executive function metrics post 12- or 24-hour call in a 12-month period.

Hypothesis: Less total sleep hours will correlate with lower scores on executive function testing (Stroop test).

Aim 2: To determine the physiologic effects of sleep deprivation from 12- and 24-hour call on heart rate variability, REM sleep, deep sleep and respiratory rate, over a 12-month period.

Hypothesis: Less total and restorative (REM and deep sleep) will correlate with lower executive function scores and higher call burden (frequency and duration) will be associated with a prolonged return to baseline in sleep metrics (total sleep, REM sleep, deep sleep, sleep consistency).

ELIGIBILITY:
Inclusion Criteria:

* Cardiology fellows at Thomas Jefferson University Hospital (PGY4-PGY6)
* Own a smart phone for Bluetooth pairing with WHOOP strap 4.0

Exclusion Criteria:

* Allergies, contraindications, or unwillingness to wear a wrist device for the study period

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiology fellows at Thomas Jefferson University Hospital (PGY4-PGY6)
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Total sleep hours per night | 180 days
  Sleep (hours per night) will be objectively measured nightly.
Executive function test (Stroop test), daily | 180 days, measured following each 24 hour call shift (weekly)
  The Stroop test demonstrates cognitive interference where a delay in the reaction time of a task occurs due to a mismatch in stimuli.
  A basic task that demonstrates this effect occurs when there is a mismatch between the name of a color (e.g. "blue" or "red") and the color it is printed on (i.e the word "red" printed in blue ink instead of red ink). When asked to name the color of the word it takes longer and is more prone to errors than when the color of the ink matches the name of the color.
  The test consists of 3 labels, each displaying the name of a color (not necessarily tinted in the color which they denote). The subject is tasked to tap on the appropriate label at the bottom, whose text denotes the ink color of the top label. The total score is the number of correct answers in 60 seconds (+1), minus the number of incorrect answers (-1). Scores may range from 0-60, with mean scores in the range of 10-20. The stroop test will be performed daily (every morning).

SECONDARY OUTCOMES:
REM sleep hours, nightly | 180 days
  REM sleep hours will be measured nightly by the WHOOP strap 4.0.
Deep sleep hours, nightly | 180 days
  Deep sleep hours will be measured nightly by the WHOOP strap 4.0.
Resting heart rate, nightly | 180 days
  Resting heart rate will be measured nightly by the WHOOP strap 4.0.
Heart rate variability, nightly | 180 days
  Heart rate variability will be measured nightly by the WHOOP strap 4.0.
Respiration rate, nightly | 180 days
  Respiration rate will be measured nightly by the WHOOP strap 4.0.
Pulse oximetry, nightly | 180 days
  Pulse oximetry will be measured nightly by the WHOOP strap 4.0.
Body temperature, nightly | 180 days
  Body temperature will be measured nightly by the WHOOP strap 4.0.
Average duty hours per week | 180 days
  Duty hours will be self-reported every week
Perceived Stress Scale-4 (PSS-4) | 180 days
  The PSS-4 consists of 4 items that assess perceived stress. The items are scored on a 4-point scale. This survey will be administered biweekly.
Patient Health Questionnaire-9 (PHQ-9) | 180 days
  The Patient Health Questionnaire-9 (PHQ-9) consists of 9 items that assess major depressive disorder. This survey will be administered biweekly. PHQ-9 score can range from 0 to 27, with 27 being most severe (worse).
Physician Well-Being Index (PWBI) | 180 days
  The Physician Well Being Index is a 7 question survey, scored 0-7, with lower scores indicative of better physician well being.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hajduczok, MD, Principal Investigator — Thomas Jefferson University Hospital, Department of Cardiology
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No